CLINICAL TRIAL: NCT00182260
Title: ELVIS (Esophagitis-Laparoscopy Versus Inhibitors of Secretion) A Randomized Controlled Trial of Laparoscopic Nissen Fundoplication (LNF) Versus Omeprazole for Treatment of Patients With Chronic Gastro-Esophageal Reflux Disease (GERD)
Brief Title: A Randomized Controlled Trial of Laparoscopic Nissen Fundoplication Treatment of Patients With Chronic GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Mehran Anvari, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR-MCT-38147; MOH Grant 05276
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Proton Pump Inhibitors

ARMS (2):
- Proton Pump Inhibitor (Active Comparator): Patients randomized to medical therapy received optimized treatment with PPI using a standardized management protocol based on best evidence and published guidelines.
  Interventions: Drug: Proton Pump Inhibitors
- Laparoscopic Nissen Fundoplication (Active Comparator): Surgical patients underwent LNF using previously published technique.
  Interventions: Procedure: Laparoscopic Nissen Fundoplication

INTERVENTIONS:
Drug: Proton Pump Inhibitors
  Arms: Proton Pump Inhibitor
Procedure: Laparoscopic Nissen Fundoplication
  Arms: Laparoscopic Nissen Fundoplication

SUMMARY:
LNF is an effective intervention in the management of patients with chronic GERD requiring maintenance therapy. LNF is cost-effective compared with long-term medical therapy.

LNF is more effective than maximum medical therapy in control of respiratory symptoms and complications of GERD.

DETAILED DESCRIPTION:
GERD encompasses a variety of symptoms and pathological findings caused by the reflux of gastric contents into the esophagus although symptoms and pathology may occur independently of each other. GERD usually presents with typical symptoms of retrosternal burning (heartburn) with or without chest pain and regurgitation of gastric contents into the back of the mouth. However, symptoms often occur in the absence of abnormalities associated with GERD, such as esophageal erosions, ulceration, stricturing or Barrett's esophagus. There is no clear correlation between symptoms and the histological features of GERD. Less prevalent manifestations of GERD include the geneses of dental erosions and respiratory disease including aspiration pneumonia, asthma, chronic laryngitis. Most often, GERD is due to excessive reflux of gastric contents into the esophagus rather than gastric acid hypersecretion. Reflux is caused by an increase in the frequency of inappropriate transient relaxations of the lower esophageal sphincter (LES). In most patients, basal resting LES pressure is normal although LES hypotonia, reduced esophageal body contractility and the presence of a hiatus hernia may exacerbate reflux or reduce esophageal clearance. Impaired esophageal mucosal resistance can increase the potential for esophageal damage. Bile acids and pancreatic enzymes have been implicated in the pathogenesis of GERD but it is generally accepted that the major causes of esophageal symptoms and injury are gastric acid and pepsin, which are active only at low ambient pH. Severity of esophagitis and of reflux symptoms correlate well with the duration of esophageal acid exposure with clear correlation between acid secretory inhibition and esophagitis healing rates for any given drug. On this basis, treatment for GERD has been directed towards:

Minimization of potential precipitating factors by lifestyle modifications such as weight loss, small meals and, avoidance of alcohol and tobacco.

Improving LES pressure, esophageal clearance and gastric emptying, using prokinetic agents.

Neutralization of acid in the stomach or esophagus, using antacids. Reduction of acid secretion, using histamine receptor antagonists(H2RAs) or PPI's.

Surgical prevention of gastro-esophageal reflux by fundoplication. In practice, the latter two approaches are the most successful for patients with more severe GERD and PPI's have proven more efficacious than H2RAs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female GERD patients aged 18-70 years with GERD symptoms.
* Prior long-term treatment with PPI with minimum duration of 1 year with expected future duration of at least 2 more years.
* Controlled on 20-40mg/day maintenance PPI therapy prior to study, defined as GERD symptom score<18 and score of 70 or more on 1-100 Global Rating Scale at screening (on medication).
* Increase in GERD symptom score>=15 points at baseline (off omeprazole).
* GERD symptom score>=18 at baseline (off omeprazole).
* Percent acid reflux in 24hr 4% at baseline (off omeprazole).
* Positive Bernstein test at baseline.
* Willingness to adhere to randomized treatment with availability for 3 years of follow-up.
* Ability to answer self and interviewer-administered questions in English.
* Signed informed consent.

Exclusion Criteria:

* Aperistaltic esophagus.
* Severe cardiac, respiratory, hematologic or other disease constituting an unacceptable surgical risk in the investigator's opinion.
* Previous gastric, esophageal or anti-reflux surgery.
* History of malignancy within the last year with the exception of basal cell carcinoma.
* Pregnancy or an intention to become pregnant in the following year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2000-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
GERD Symptom Scale
Symptom-free Day Measurement
Cost Measurement

SECONDARY OUTCOMES:
24-hour pH
Economic Analysis
Endoscopy
Esophageal manometry
Health related quality of life (SF-36)
Health Utility Index
Respiratory function, airways hypersensitivity and inflammation and microaspiration

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Anvari, MB, BS, PhD, Principal Investigator — McMaster University; David Armstrong, MB, BCh, MA, Principal Investigator — McMaster University; Charles H. Goldsmith, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada